CLINICAL TRIAL: NCT07141043
Title: New Directions and Perspectives in the Assessment of Mineral and Bone Disorders in Kidney Transplant Recipients
Brief Title: Assessment of Mineral and Bone Disorders in Kidney Transplant Recipients
Status: Recruiting | Type: Observational
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Akad Nada, MD, Grigore T. Popa University of Medicine and Pharmacy
Other Study IDs: Nr. 501/30.11.2024
Record Dates: First submitted 2025-06-28; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Hemodyalysis; Kidney Tansplant; Osteoporosis; CKD-MBD - Chronic Kidney Disease Mineral and Bone Disorder
Keywords: CKD-MBD; Osteoporosis; bone turnover markers
MeSH Terms: conditions — Osteoporosis; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hemodialysis group: Patients undergoing HD for at least 12 months, aged 20-70 years, after signing an informed consent.
- Kidney transplant group: Patients with successful KTx performed at least 12 months prior to their enrollment, aged 20-70 years old, after signing an informed consent. Subjects will be eligible for inclusion regardless of KTx immunosuppression regimen, pre-transplantation history, history of pre-transplant dialysis, or whether the kidney donation was from a living or deceased donor.
- General population osteoporosis/osteopenia: Men and postmenopausal women diagnosed with primary osteopenia or osteoporosis, aged 50-70 years old, after signing an informed consent.

SUMMARY:
This study aims to integrate bone measurements (including bone turnover markers (BTM), bone mineral density (BMD) measurement, vertebral fracture assessment (VFA), trabecular bone score (TBS) ) commonly used in the general population for primary osteoporosis evaluation to enhance the assessment of CKD-MBD.

DETAILED DESCRIPTION:
Prospective observational study that will evaluate differences in bone (BMD, TBS, VFA and BTMs, serum calcium and phosphate) parameters in hemodialysis (HD) patients and kidney transplant recipients (KTR), compared to general population osteopenia/osteoporosis patients, at baseline and after one year of monitoring, with or without therapeutic intervention for CKD-MBD (KTR and HD groups).

ELIGIBILITY:
Inclusion Criteria:

1. HD group: Patients undergoing HD for at least 12 months, aged 20-70 years, after signing an informed consent.
2. KTR group: Patients with successful KTx performed at least 12 months prior to their enrollment, aged 20-70 years old, after signing an informed consent. Subjects will be eligible for inclusion regardless of KTx immunosuppression regimen, pre-transplantation history, history of pre-transplant dialysis, or whether the kidney donation was from a living or deceased donor.
3. GPO group: men and postmenopausal women diagnosed with primary osteopenia or osteoporosis, aged 50-70 years old, after signing an informed consent.

Exclusion Criteria:

1. HD group: Treatment with active bone therapies (excluding calcium and vitamin D); ongoing cancer treatment or recent history of malignancy, cirrhosis, recent major fractures, patients who have received transplants other than kidney, secondary causes of osteoporosis (other than CKD or transplant-related: primary hyperparathyroidism, hyperthyroidism, congenital bone disorders, sarcoidosis, severe bone trauma, malignant tumors, inflammatory bowel disease, endogenous Cushing syndrome, anti-estrogen/anti-androgen therapy, and anorexia nervosa), pregnancy and breast-feeding.
2. KTR group: The same as for HD + return to dialysis + acute graft rejection.
3. GPO group: The same as for HD + diabetes mellitus + prolonged glucocorticoid therapy (>7.5 mg Prednisone or equivalent for at least 3 months).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and postmenopausal women diagnosed with primary osteopenia or osteoporosis, aged 50-70 years old and patients undergoing HD or KTR, aged 20-70 years old.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in BTM Levels in KTx recipients (KTR) compared to HD patients and general population osteopenia/osteoporosis (GPO) patients. | 12 months
  Longitudinal assessment of BTMs, including serum procollagen type I N-terminal propeptide (P1NP), osteocalcin, bone specific alkaline phosphatase (BAP), C-terminal telopeptide of type I collagen (CTX) and tartrate-resistant acid phosphatase 5b (TRAP5b) in KTR compared with HD patients and GPO patients.

SECONDARY OUTCOMES:
Correlation Between BTM Levels and BMD in KTR compared with HD and GPO patients. | 12 months
  Correlation analysis between BTM levels (procollagen type I N-terminal propeptide (P1NP), osteocalcin, bone specific alkaline phosphatase (BAP), C-terminal telopeptide of type I collagen (CTX) and tartrate-resistant acid phosphatase 5b (TRAP5b)) and BMD (g/cm²) assessed by dual-energy X-ray absorptiometry (DXA) at the lumbar spine, femoral neck and forearm. Data will be stratified by study group (KTR, HD and GPO patients) and by gender. Correlation coefficients will be reported for each group.
Correlation Between BTM Levels and TBS in KTR compared with HD and GPO patients. | 12 months
  Correlation analysis between BTM levels (procollagen type I N-terminal propeptide (P1NP), osteocalcin, bone specific alkaline phosphatase (BAP), C-terminal telopeptide of type I collagen (CTX) and tartrate-resistant acid phosphatase 5b (TRAP5b)) and TBS (unitless index) derived from DXA images at the lumbar spine. Data will be stratified by study group (KTR, HD and GPO patients) and by gender. Correlation coefficients will be reported for each group.
Key BTMs Predicting Bone Health Outcomes in KTR Patients | 12 months
  Correlation between change from baseline in BTM and change from baseline in TBS.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medicine and Pharmacy "Grigore T. Popa", Iași, Romania

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy concerns and data protection regulations.